CLINICAL TRIAL: NCT07257211
Title: Unicompartimental vs Total Knee Arthroplasty for Medial Knee Osteoarthritis: a Prospective, Ramdomized, Controlled Study
Brief Title: Partial vs Total Knee Replacement for Medial Knee Osteoarthritis: a Prospective Randomized Controlled Study
Acronym: UKA vs TKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1404/2025
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Medial Knee Osteoarthritis
Keywords: unicompartmental; knee arthroplasty; partial knee replacement; total knee replacement; randomized controlled trial; knee prosthesis
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UKA (Active Comparator): patients receiving a unicompartmental knee arthroplasty
  Interventions: Procedure: unicompartmental knee arthroplasty
- TKA (Active Comparator): patients receiving a total knee arthroplasty
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: unicompartmental knee arthroplasty — medial unicompartmental knee arthroplasty using standard surgical technique and routine postoperative care
  Arms: UKA
Procedure: total knee arthroplasty — total knee arthroplasty using standard surgical technique and routine postoperative care
  Arms: TKA

SUMMARY:
The goal of this clinical trial is to learn whether partial knee replacement (unicompartmental knee arthroplasty, UKA) or total knee replacement (total knee arthroplasty, TKA) leads to better clinical and functional outcomes in adults with medial knee osteoarthritis who are candidates for knee arthroplasty.

The main questions the study aims to answer are:

* Does UKA or TKA result in better patient-reported outcomes, such as knee pain, function, and quality of life (measured by Oxford Knee Score, WOMAC, and Knee Society Score)?
* Does UKA or TKA lead to differences in complications or revision rates during follow-up?

Researchers will compare UKA to TKA to see whether one procedure provides superior postoperative recovery, knee function, and long-term outcomes under standard clinical care conditions.

Participants will:

* Receive either a unicompartmental or total knee replacement, assigned by randomization.
* Undergo routine postoperative examinations, including standardized questionnaires (e.g., Oxford Knee Score, WOMAC, Knee Society Score, VAS).
* Attend follow-up visits at standard clinical intervals (e.g., 6 weeks, 6 months, 1 year, 2 years, and beyond).

DETAILED DESCRIPTION:
Medial knee osteoarthritis is a common degenerative joint disease that often leads to significant pain, loss of function, and reduced quality of life. When conservative treatments are no longer effective, surgical joint replacement is a standard therapeutic option. Two established procedures are unicompartmental knee arthroplasty (UKA), which replaces the diseased medial compartment, and total knee arthroplasty (TKA). Both procedures are widely used, but it remains unclear which option provides better outcomes for patients who specifically present with isolated medial osteoarthritis.

This prospective, randomized, controlled clinical trial aims to systematically compare the functional, radiological, and patient-reported outcomes of UKA and TKA performed under routine clinical care conditions. The study is conducted at the Department of Orthopaedics and Traumatology at the Medical University of Graz. Adult patients with isolated medial knee osteoarthritis who meet established clinical and radiographic criteria for knee arthroplasty are eligible for participation.

All surgical procedures are performed using standard techniques and implants currently approved and used in routine practice. Postoperative follow-up follows the usual clinical schedule (e.g., 6 weeks, 6 months, 1 year, 2 years), with additional long-term clinical and radiological assessments as part of institutional standard care. During these visits, participants complete validated patient-reported outcome measures, including the Oxford Knee Score, WOMAC, Knee Society Score, Forgotten Joint Score, and Visual Analog Scale for pain. Radiographs are collected to assess implant position and alignment.

The study seeks to determine whether one of the two surgical approaches results in superior knee function, less postoperative pain, faster recovery, or lower complication and revision rates. Findings from this trial may support evidence-based decision-making for surgeons and patients considering knee arthroplasty for isolated medial knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* written consent, 4th degree medial osteoarthritis, max 1st degree lateral osteoarthritis, max. 2nd degree osteoarthritis in patellofemoral joint

Exclusion Criteria:

* from 2nd degree lateral osteoarthritis, from 3nd degree osteoarthritis in patellofemoral joint, non-compensatable varus or valgus misalignment above 10 degrees, non-consent, age under 40 / over 90, st.p. fracture of the femur and or tibi, infection, st.p. joint replacement or osteotomy in the area of the knee joint, simultaneus bilateral care, pregnany

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
clinical functional outcome (KOOS) | 12 months
  KOOS evaluates patient reported knee function, pain, symptoms, activities of daily living, and quality of life. Higher score indicates better outcomes.

SECONDARY OUTCOMES:
complication rate within 12 months | 12 months
  include infection, thromboembolic events, reintervention, and other adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Department for orthopedics and traumatology of Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided